CLINICAL TRIAL: NCT00505531
Title: Pain Study to See if Ultram ER Will Provide Relief to Subjects Whose Pain is Not Well Controlled by Narcotics
Status: Terminated | Type: Observational
Why Stopped: Not enough data to analyze the results.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Ortho-McNeil, Inc. (Industry)
Responsible Party: Principal Investigator, Jianren Mao, MD, PhD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2007P 000025
Record Dates: First submitted 2007-07-19; First posted 2007-07-23 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Chronic Pain
Keywords: Pain
MeSH Terms: conditions — Chronic Pain; Pain | interventions — Tramadol; Diphenhydramine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Tramadol ER- 200mg: Tramadol Extended Release capsules Weeks 1 & 6- 100 mg/day Weeks 2-5- 200 mg/day
  Interventions: Drug: Tramadol Extended Release Oral Capsule
- Tramadol ER- 300mg: Tramadol Extended Release capsules Weeks 1 & 7- 100 mg/day Weeks 2 & 6- 200 mg/day Weeks 3-5- 300 mg/day
  Interventions: Drug: Tramadol Extended Release Oral Capsule
- Placebo: Diphenhydramine capsules Weeks 1-6- 25 mg/day
  Interventions: Drug: Benadryl

INTERVENTIONS:
Drug: Tramadol Extended Release Oral Capsule — Tramadol ER- up to either 200 mg or 300 mg based on randomization
  Other Names: Ultram ER
  Groups: Tramadol ER- 200mg; Tramadol ER- 300mg
Drug: Benadryl — Placebo group will take up to 25 mg of Benadryl
  Other Names: Diphenhydramine
  Groups: Placebo

SUMMARY:
The Massachusetts General Hospital Center for Translational Pain Research is conducting a research study to see if Ultram ER, an FDA-approved pain medication, would be helpful in providing pain relief in subjects whose chronic pain is not well controlled on narcotic pain medicine.

DETAILED DESCRIPTION:
The study consists of 6 visits over 6 weeks. Study testing includes: physical exam, urine testing, questionnaires and non-invasive (no needles) nerve testing using cold/heat sensations. Compensation and some parking reimbursement provided.

ELIGIBILITY:
Inclusion Criteria:

1. Subject will be between ages 18 to 65 years in all three groups.
2. Subject has NOT been on Tramadol or Tramadol ER for at least one month.
3. Subject has NOT been on tricyclic antidepressants, serotonin, norepinephrine, or mixed serotonin/norepinephrine reuptake inhibitors (SSRI/SNRI), or muscle relaxant with potential action as an SSRI or SNRI (e.g., Flexeril) for at least one month. Subject has not been on monoamine oxidase inhibitors in the past 14 days.
4. Subjects should have had a stable pain condition (e.g., axial low back pain as listed below in item # 5-7) for at least three months. This requirement is set in order to avoid clinical uncertainty from an unstable pain condition and to minimize the study variation.
5. Axial low back pain refers to pain conditions resulting from myofascial disorder, lumbar facet joint disease, discogenic disease, and postlaminectomy syndrome. Patients with neurological signs (weakness or numbness) will not be included in the study because of potential confounding effects on the QST assessment of pain threshold and pain tolerance.
6. Headaches refer to migraine, tension, or cluster headache, cervicogenic pain (e.g., facet joint disease, myofascial pain), and trigeminal neuralgia. However, patients with neurological diseases including multiple sclerosis, amyotrophic lateral sclerosis, and stroke will not be included due to possible neurological deficits that may confound the QST assessment.
7. Abdominal and pelvic pain refers to pain from abdominal and/or pelvic organs (e.g., chronic pancreatitis, endometriosis).
8. Subject is willing to have his/her opioid dose tapered.
9. Female subjects of childbearing potential must have a negative urine pregnancy test at the initial visit.

Exclusion Criteria:

1. Subject has sensory deficits at the sites of QST. Sensory deficits refer to such changes resulting from neurological diseases or medical conditions causing peripheral polyneuropathy and sensory changes, which include but are not limited to diabetes, alcoholic neuropathy, AIDS neuropathy, thyroid disease, severe liver or kidney disorders.
2. Subject has scar tissue, infection, or acute injury at the sites of QST.
3. Subject has had interventional procedures that may alter the results of QST. Such procedures include neuroablation (chemical or electrothermal) at any time, neuraxial (e.g., epidural) or local anesthetic block within the last eight weeks, and lumbar sympathetic or hypogastric block within the last six months. We consider eight weeks and six months as the minimal time period that must have elapsed after neuraxial injection and lumbar sympathetic block, respectively, in order to minimize the possible influence from a previous interventional procedure.
4. Subject has a pending litigation related to his/her chronic pain condition.
5. Subject has a history of or current seizure disorder.
6. Subject has a history of severe allergic reaction to Tramadol ER or other opioid medications.
7. Subject has a major psychiatric disorder (major depression; bipolar disorder; schizophrenia; anxiety disorder; psychotic disorders; eating disorders; alcohol or drug dependence; attention deficit hyperactivity disorder); subject with any known history of such conditions also will be excluded.
8. Subject has severe renal impairment or severe hepatic impairment.
9. Subject is using illicit drugs detected through the urine toxicology screen.
10. Subject is pregnant or lactating.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects whose chronic pain is not well controlled on narcotic pain medicine.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Tramadol ER reduces VAS for patients with OIH | 6 weeks
  VAS will be recorded at each visit and then analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Jianren Mao, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Center for Translational Pain Research, Boston, Massachusetts, United States